CLINICAL TRIAL: NCT02096094
Title: A Double-blind Evaluation of Adverse Effects of Bath With Wipes Impregnated With 2% Chlorhexidine Versus Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: G70 antisepsis (Unknown)
Responsible Party: Principal Investigator, Alejandro E. Macias, MD, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GTSSA002101245
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2014-03

CONDITIONS: Bed Bathing
Keywords: Antiseptics; Administration cutaneously; Chlorine compounds; Infection control; Anti-infecting agents, local
MeSH Terms: interventions — Baths; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine bath (Experimental): This arm is composed with 27 healthy volunteers which will perform full body bath with wipes impregnated with 2% chlorhexidine and with shampoo with 0.15% chlorhexidine.
  Interventions: Procedure: Standardization phase; Procedure: Bath with chlorhexidine
- Control bath (Placebo Comparator): This arm is composed with 27 healthy volunteers which will perform full body bath with wipes and shampoo without chlorhexidine.
  Interventions: Procedure: Standardization phase; Procedure: Control bath

INTERVENTIONS:
Procedure: Standardization phase — Prior the principal intervention, each volunteer should complete a standardization phase, which consists in the daily bathing for two weeks with a antiseptic free soap and shampoo. Likewise would avoid chemical showers such as swimming. At the end of this phase a quantification of skin flora will be perform.
  Other Names: Skin flora standarization
Procedure: Control bath — Volunteers will be ask to perform full body bath with wipes without impregnation for 3 to 5 days, each day the volunteer will answer a survey regarding side effects (skin reactions) and comfort related to the bath. At the end of the intervention, a skin culture to quantify skin colonization will be performed.
  Arms: Control bath
Procedure: Bath with chlorhexidine — Volunteers will be asked to perform full body bath with wipes with 2% chlorhexidine impregnation and with 0.15% chlorhexidine shampoo (for the head and genitalia) for 3 to 5 days. Each day the volunteer will answer a survey regarding side effects (skin reactions) and comfort related to the bath. At the end of the intervention, a skin culture to quantify skin colonization will be performed.
  Arms: Chlorhexidine bath

SUMMARY:
Traditional bed bathing have been related to cross-infection. In order to avoid this complication, single-use products such as wipes impregnated with chlorhexidine use is increasing. Nevertheless among nursery staff concern about its side effects prevents its widespread use. The investigators want to know if there are any differences between the use of 2% chlorhexidine wipes and a placebo concerning side effects.

DETAILED DESCRIPTION:
Hygiene is part of health recovery in patients, nevertheless in unconscious or sedated patients this procedure becomes a task for the nursing staff. Traditional soap and water bed bath is becoming obsolete as soap could induce skin injuries due to changes in the pH of the skin and furthermore, almost every items used for this procedure could be a reservoir for pathogens, and therefore could lead to infection. Nowadays single-use products are a new option for prevent cross-infections. Nevertheless, traditional bed bathing is a tightly established practice among nursing staff. New evidence about side effects and comfort by wipe bed bathing is needed.

Chlorhexidine impregnated wipes have been used to perform the bed bathing in severe ill patients, as it can protect them from infections. The aim of this study is to determinate if bed bathing with 2% chlorhexidine impregnated wipes has a similar effect that a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteer

Exclusion Criteria:

* History of skin allergies or atopy, as well as reactions to soaps or chlorine compounds.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Skin reaction to chlorhexidine | 24 hours
  Presence of any cutaneous reaction in the first 24 hours after bathing with chlorhexidine. If the volunteers develop any skin reaction, a blinded dermatologist will evaluate it, and will perform a susceptibility test to determine if skin reaction is related to the antiseptic.

SECONDARY OUTCOMES:
Comparison of bacterial colony count of skin. | 24 hours
  Comparison of bacterial colony counts of skin after and before the intervention. After incubation, a blinded technician will count the colonies to determine the colony-forming units per square centimeter (CFU/cm2) of skin for each bacterial colony count.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro E Macias, MD, Principal Investigator — Universidad de Guanajuato; Juan L Mosqueda, MD, Study Director — Universidad de Guanajuato; Ruth C Morales, MD, Study Chair — Universidad de Guanajuato; Virginia Arreguin, MD, Study Chair — Universidad de Guanajuato; Jose A Alvarez, MD, Study Chair — Universidad de Guanajuato; Juan M Munoz, MD, Study Chair — Universidad de Guanajuato; Juan H Macias, MD, Study Chair — Universidad de Guanajuato
Locations (1):
- General Hospital of Leon, León, Guanajuato, Mexico